CLINICAL TRIAL: NCT00640068
Title: Advanced Cardiovascular Imaging Consortium: A Collaborative Quality Improvement Project
Brief Title: Advanced Cardiovascular Imaging Consortium
Acronym: ACIC
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Kavitha Chinnaiyan, Medical Director of Noninvasive Cardiology Education; Program Director, ACIC, Corewell Health East
Other Study IDs: 2007-236
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Chest Pain; Coronary Occlusion; Coronary Artery Disease
Keywords: coronary artery disease; chest pain; coronary artery bypass graft; stress test; Coronary Angiography
MeSH Terms: conditions — Chest Pain; Coronary Occlusion; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All patients in whom a clinical CCTA was ordered by their physician at a participating site. Patient must have a prescription for CCTA ordered by their physician.

SUMMARY:
The ACIC is a Collaborative Quality Improvement (CQI) program involving the collection of data related to: indications for Coronary Computed Tomography (CCTA), patient health characteristics, acquisition techniques of CCTA scans, physician interpretation of results and short-term outcomes over a 90 day period.

DETAILED DESCRIPTION:
This study is a collaborative quality assurance initiative organized by Blue Cross Blue Shield of Michigan and Blue Cross Network (BCBSM/BCN) for initiation of insurance coverage of coronary artery CT scanning (CCTA), a relatively new procedure that can provide non-invasive coronary angiograms. While this procedure has promise in that it can rapidly diagnose patients with unknown chest pain and reduce the cost of medical care, there is substantial potential for abuse and excess cost and inappropriate care if not appropriately used.

The Consortium's objectives are to educate participating sites of the clinical uses of CCTA as well as other best-practice recommendations; to create a database (Registry) to develop evidence of the best-practice utilization of CCTA; to provide a feedback mechanism to the sites about the positive or negative evidence of best-practice utilization of CCTA; to develop strategies to improve the utilization of CCTA; to monitor the CQI process of the individual participating sites; to reduce cost and improve safety and efficiency in in the care of patients with acute chest pain, indeterminate stress tests results, and to assess coronary bypass graft patency.

ELIGIBILITY:
Inclusion Criteria:

(Patient must meet one criteria)

* Patient has had a CCTA examination ordered by a referring physician at a participating site.
* Patient is a self referral.

Exclusion Criteria:

Clinical contraindications to CCTA are present as determined by attending physician or staff, including but not limited to:

* Pregnancy or potential pregnancy.
* Renal failure or dysfunction.
* Inability to receive beta blockers.
* Allergy to iodinated contrast without prior premedication.
* Unwillingness to participate.
* Inability to read or understand Patient Information Sheet.
* Age less than 18 years without parent or guardian's evaluation of Patient Information Sheet. Underage and other vulnerable populations are included as the CQI process is intended to detect and correct adverse consequences of CCTA, e.g., excessive radiation, and protect such patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Referral from other healthcare provider or support staff (e.g. physician office, clinics), Emergency Room, self referral with prescription
Sampling Method: Non-Probability Sample
Enrollment: 42926 (Actual)
Dates: Start 2007-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Educate participating sites on appropriate use of CCTA | 5 years
  To educate participating sites in the clinical uses of CCTA recommended by the ACC/ACR as well as other best-practices

SECONDARY OUTCOMES:
To monitor the CQI process of individual participating sites and the ACIC as a whole. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Chinnaiyan, MD, Study Director — Corewell Health East
Locations (50):
- United States (50):
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - DMC Huron Valley-Sinai, Commerce, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Premier Medical Clinics, Flint, Michigan
  - Garden City Hospital, Garden City, Michigan
  - North Ottawa Community Hospital, Grand Haven, Michigan
  - East Beltline Imaging, Grand Rapids, Michigan
  - Henry Ford Cottage Hospital, Grosse Pointe, Michigan
  - William Beaumont Hospital - Grosse Pointe, Grosse Pointe, Michigan
  - Hillsdale Community Health Center, Hillsdale, Michigan
  - Bronson Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Health System, Lansing, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Thoracic and Cardiovascular Institute, P.C., Lansing, Michigan
  - McLaren Lapeer Region, Lapeer, Michigan
  - St. John Oakland, Madison Heights, Michigan
  - Marquette General Health System, Marquette, Michigan
  - Mercy Memorial, Monroe, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Pontiac Osteopathic Hospital, Pontiac, Michigan
  - St. Joseph Mercy Hospital Oakland, Pontiac, Michigan
  - Crittenton Hospital, Rochester, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Covenant Healthcare, Saginaw, Michigan
  - Lakeland Regional Health System, Saint Joseph, Michigan
  - Chippewa County War Memorial, Sault Saint Marie, Michigan
  - St. John Providence Hospital, Southfield, Michigan
  - Southgate Radiology & Southgate CT, Southgate, Michigan
  - St. Joseph Health System - Tawas, Tawas City, Michigan
  - Heritage (Oakwood) Hospital, Taylor, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Oakwood Southshore Medical Center, Trenton, Michigan
  - William Beaumont Hospital, Troy, Troy, Michigan
  - St. John Macomb, Warren, Michigan
  - Oakwood Annapolis Hospital, Wayne, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Health First Imaging, West Bloomfield, Michigan
  - West Branch Regional Medical Center, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Michigan Heart, P.C., Ypsilanti, Michigan

REFERENCES:
- [Derived] Burris AC 2nd, Boura JA, Raff GL, Chinnaiyan KM. Triple Rule Out Versus Coronary CT Angiography in Patients With Acute Chest Pain: Results From the ACIC Consortium. JACC Cardiovasc Imaging. 2015 Jul;8(7):817-25. doi: 10.1016/j.jcmg.2015.02.023. Epub 2015 Jun 17. PMID 26093928
- [Derived] Chinnaiyan KM, Boura JA, DePetris A, Gentry R, Abidov A, Share DA, Raff GL; Advanced Cardiovascular Imaging Consortium Coinvestigators. Progressive radiation dose reduction from coronary computed tomography angiography in a statewide collaborative quality improvement program: results from the Advanced Cardiovascular Imaging Consortium. Circ Cardiovasc Imaging. 2013 Sep;6(5):646-54. doi: 10.1161/CIRCIMAGING.112.000237. Epub 2013 Aug 7. PMID 23926193
- [Derived] Chinnaiyan KM, Depetris AM, Al-Mallah M, Abidov A, Ananthasubramaniam K, Gallagher MJ, Girard S, Goraya TY, Kazerooni EA, Patel S, Peyser P, Poopat C, Raff GL, Saba S, Song T, Share D. Rationale, design, and goals of the Advanced Cardiovascular Imaging Consortium (ACIC): A Blue Cross Blue Shield of Michigan collaborative quality improvement project. Am Heart J. 2012 Mar;163(3):346-53. doi: 10.1016/j.ahj.2011.11.018. PMID 22424004
- [Derived] Chinnaiyan KM, Raff GL, Goraya T, Ananthasubramaniam K, Gallagher MJ, Abidov A, Boura JA, Share D, Peyser PA. Coronary computed tomography angiography after stress testing: results from a multicenter, statewide registry, ACIC (Advanced Cardiovascular Imaging Consortium). J Am Coll Cardiol. 2012 Feb 14;59(7):688-95. doi: 10.1016/j.jacc.2011.10.886. PMID 22322086
- [Derived] Vanhecke TE, Madder RD, Weber JE, Bielak LF, Peyser PA, Chinnaiyan KM. Development and validation of a predictive screening tool for uninterpretable coronary CT angiography results. Circ Cardiovasc Imaging. 2011 Sep;4(5):490-7. doi: 10.1161/CIRCIMAGING.111.964205. Epub 2011 Jul 20. PMID 21775504
- [Derived] Raff GL, Chinnaiyan KM, Share DA, Goraya TY, Kazerooni EA, Moscucci M, Gentry RE, Abidov A; Advanced Cardiovascular Imaging Consortium Co-Investigators. Radiation dose from cardiac computed tomography before and after implementation of radiation dose-reduction techniques. JAMA. 2009 Jun 10;301(22):2340-8. doi: 10.1001/jama.2009.814. PMID 19509381